CLINICAL TRIAL: NCT07011901
Title: Dissecting Neurocognitive Components of Compulsivity Using Computational Modeling and EEG
Brief Title: Precision Analytic Research Methods in OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amy Rapp, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-01125; K23MH133997 (NIH)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Obsessive Compulsive Disorder; Exposure and response prevention; Cognitive Behavioral Therapy; Electroencephalogram
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants diagnosed with OCD (Experimental): All participants diagnosed with Obsessive Compulsive Disorder (OCD) who enroll in this study will receive 17 sessions of exposure and response prevention, a specialized cognitive behavioral therapy for OCD, over the course of 10 weeks.
  Interventions: Behavioral: Exposure and Response Prevention
- Healthy controls (No Intervention): Individuals who do not have a current or lifetime psychiatric diagnosis will not receive any treatment.

INTERVENTIONS:
Behavioral: Exposure and Response Prevention — Exposure and response prevention (EX/RP) is the gold-standard behavioral treatment for OCD. It involves confronting the content of obsessions (distressing thoughts, images, or impulses) and resisting the urge to engage in compulsions (observable behaviors or mental acts that are repeated to reduce the anxiety/distress associated with compulsions).
  Arms: Participants diagnosed with OCD

SUMMARY:
Psychiatric disorders characterized by compulsivity, such as obsessive-compulsive disorder (OCD), result in considerable functional impairment and many individuals do not respond to gold-standard treatments. Compulsivity has long been thought to occur due to exaggerated habits and reduced goal-directed control, although more recently, this conceptualization of compulsivity as an imbalance of two cognitive systems has been challenged as overly narrow. This study will recruit 100 individuals (50 adults diagnosed with OCD, 50 healthy controls) and leverage the measurement precision offered by theory-driven computational modeling in combination with electroencephalogram (EEG) to go beyond this binary theory of compulsivity, revealing how more complex interactions of neurocognitive subcomponents contribute to compulsivity-information that could ultimately lead to improved treatment personalization and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Participants must be:

* between the ages 18-55 years old
* English-speaking
* right-handed
* able to provide consent

Exclusion Criteria:

Individuals diagnosed with OCD will be excluded if:

* they meet diagnostic criteria for certain other psychiatric disorders
* are taking psychiatric medication or have received behavioral treatment for OCD within a certain timeframe
* if it is unsafe for them to participate in research

Healthy control participants will be excluded if:

* they have a current psychiatric disorder
* a lifetime history of certain psychiatric disorders
* are taking psychiatric medication or have in the past
* have a parent or sibling who has been diagnosed with OCD
* if it is unsafe for them to participate in research

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | Week 1, Week 5, Week 10
  A semi-structured clinician-administered instrument used to measure obsessions and compulsions separately over five dimensions (time consumed, distress, interference, degree of resistance, control). The range of scores for the Obsessions and Compulsions subscales is 0-20, and the range for the total score is 0-40. Higher scores indicate greater symptom severity, and a total score greater or equal to 16 is considered indicative of moderately severe OCD

SECONDARY OUTCOMES:
Obsessive Compulsive Inventory- Revised | Week 1, Week 5, Week 10
  An 18-item self-report measure to assess obsessions and compulsions that demonstrates good psychometric properties and has been used in other research as a transdiagnostic measure of compulsivity. The range of scores for the six subscales (Washing; Obsessing; Ordering; Checking; Neutralizing; Hoarding) is 0-12. The range for the total score is 0-60 and does not include the Hoarding subscale. Higher scores indicate greater symptom severity.
Cambridge-Chicago Compulsivity Trait Scale | Week 1, Week 5, Week 10
  A 15-item self-report measure to assess compulsivity transdiagnostically that exhibits high internal consistency and excellent convergent validity with gold-standard measures of compulsive symptoms. The range for the total score is 0-45, with higher scores indicating greater symptom severity
Self-Report Habit Index | Week 1, Week 5, Week 10
  A 12-item self-report measure of the repetition and automaticity of a behavior that exhibits high internal consistency and test-retest reliability. The range for the total score is 12-84, with higher scores indicating greater symptom severity.
Dimensional Obsessive- Compulsive Scale | Week 1, Week 5, Week 10
  A 20-item self-report measure that assesses four of the most consistently replicated thematic dimensions of OCD symptoms (i.e., contamination, harm, symmetry, repugnant content). The DOCS demonstrates good to excellent internal consistency, validity, and sensitivity. The range of scores for the four subscales (Contamination; Harm; Unacceptable Thoughts; Symmetry) is 0-20, and the range for the total score is 0-80. Higher scores indicate greater symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Rapp, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Analytic Code
Time Frame: Deidentified data will be deposited to the Open Science Framework (OSF) and the NIMH Data Archive (NDA), in line with data sharing requirements stipulated by the NIMH. In addition to the patient level data, experimental task design specifications will be shared to OSF and posted on the Principal Investigator's (Amy Rapp) GitHub page. A data dictionary will be uploaded to the NDA. Researchers who are interested in obtaining data from this study to submit a written request which would allow access for one year and would be renewable. Deidentified data will be stored indefinitely in the NDA.
Access Criteria: Researchers who provide a methodologically sound proposal will be given access to deindentified study data needed to achieve aims in the approved proposal. Data will be available indefinitely at site link (to be determined).